CLINICAL TRIAL: NCT06519539
Title: Implementing Strategies for Eating Behaviour Modification Based on Portion Control: Methodological Development and Pilot Study
Brief Title: Implementing Strategies for Eating Behaviour Modification Based on Portion Control
Acronym: PORTIONS-4
Status: Active, not recruiting | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: PC139-140
Record Dates: First submitted 2024-05-16; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-05

CONDITIONS: Lifestyle, Healthy; Weight Management; Behavior Change
Keywords: Portion size; Portion control tool; Dietary energy density

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with overweight or obesity: Healthy adults with a BMI of 27.5 kg/sq-m or above (26 or above for those of Asian descent), who will undertake a 6 month lifestyle intervention focused on improving dieary choices, physical activity and attitudes towards weight management.
  Interventions: Behavioral: PORTIONS-4 behaviour change strategies

INTERVENTIONS:
Behavioral: PORTIONS-4 behaviour change strategies — The intervention includes 4 components, including: a portion control tool set previously developed and tested in our laboratory; a supporting guide (physical book) with dietary, activity and behavioural recommendations; a mobile application aligned with the guide; and biweekly telephone calls from the psychologist and/or dietitian.

SUMMARY:
This is a pre-post intervention study designed to evaluate the feasibility of a self-applied weight management intervention based on portion control. A total of 40 healthy volunteers with overweight/obesity will take part in a 6-month intervention featuring 4 components: a portion control toolset; a manual including instructions for the use of the tools, dietary and activity recommendations, and behavioural strategies; a mobile app to motivate intervention engagement; and biweekly telephone support. The primary outcome will be Intervention adherence, assessed as the change in dietary energy density, meal nutrient composition and utilization of intervention components from start to end of trial. Other measurements (at baseline, 3 and 6 months from baseline) will include body composition, fasting biochemical parameters, inhibitory control, eating behaviour, portions size norms and acceptance of the intervention.

DETAILED DESCRIPTION:
According to recent meta-analyses, portion control tools represent an acceptable and potentially effective strategy to aid in weight loss. However, how well these tools work depends on their consistent use and a good integration with other lifestyle modification strategies around body weight control and overall health. The present pilot study was designed to evaluate the feasibility of a self-applied weight management intervention based on portion control and to identify factors influencing adherence. The sample will consist of 40 healthy volunteers with overweight/obesity who will engage in a pre-post intervetion study lasting six-months. The intervetion will include four components: (1) a portion control toolkit (serving spoon and oil dispenser); (2) a phsyical manual with instructions for using the tools, dietary and physical activity recommendations, and strategies to build habits and improve mental wellbeing; (3) a mobile app to motivate intervention engagement; and (4) biweekly short telephone support. Adherence to the intervention will be the primary outcome, assessed on a fortnightly basis as the change from baseline in dietary energy density and change in meal nutrient composition plus frequency of using the intervention components. Other measurements that will be taken at baseline, 3 and 6 months from baseline, will be: body composition, fasting biochemical parameters, inhibitory control (only baseline and 6 months), eating behaviour, portion size norms and intervention acceptance. After 3 months of taking part in the intervention, a subset of the sample will participate in a nominal group session aimed at identifying barriers to intervention adherence and strategies to overcome them. The study results will inform the design of a full-scale controlled trial featuring the most successful components.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index equal or above 27.5 kg/m2 (26.0 kg/m2 for those of Asian descent)
* Eating home-made meals at least 5 days a week
* Physically and mentally fit as assessed by the study researcher
* On-going pharmacological and hormonal treatment is accepted when this does not affect the study parameters (e.g. glucose response, appetite), and when the participant has been in a stable dose for at least 3 months
* Agreeing to undergo all the study procedures
* Being able to attend in person on 3 clinical investigation days during working hours
* Being able to understand and agree to sign the informed consent form

Exclusion Criteria:

* Being a regular smoker (that is, smoke more than 4 cigarettes a month)
* Being pregnant, breastfeeding or planning a pregnancy
* Exceed the alcohol consumption limit marked for the corresponding sex (more than 14 units in women and 20 units in men)
* Having followed a meal plan for weight loss and/or muscle mass gain in the 3 months prior to the start of the study intervention
* Having used a portion measuring instrument (e.g. scale, calibrated plate, etc.) consistently (at least in one main meal for at least 5 days a week) during the 3 months prior to the start of the study intervention
* Experiencing a weight change greater than 5% in the last 3 months
* History of relevant functional or structural anomalies of the digestive system, such as malformations, angiodysplasias, active peptic ulcers, chronic inflammatory or malabsorption diseases, or history of intestinal or bariatric surgery
* Suffer from some type of cancer, currently undergoing treatment for cancer, or when a period of at least 5 years has not elapsed since its eradication
* On-going chronic metabolic disease or obesity-related disease, or any systemic intestinal, liver or kidney disease such as type 1 or type 2 diabetes, severe dyslipidemia, uncontrolled thyroid function disorder, cirrhosis, inflammatory bowel disease, untreated anemia, etc. . (will not be excluded due to "fatty liver")
* Avoiding, being allergic, or being intolerant to the study foods or their ingredients (lactose free and regular chocolate milkshake)
* History of anaphylactic reaction to any food
* Taking any nutritional supplementation as a prescription medication that may affect the results of the study
* Taking over-the-counter nutritional supplementation (that is, without a medical prescription) that may affect the results of the study, unless the person is willing to stop it during the 6 months of the study duration and only when a minimum washout period of 14 days can be guaranteed prior to the basal measurements being taken
* A high incidence of attitudes and behaviors associated with eating disorders, expressed as a score greater than 20 on the 26-item Eating Attitudes Test scale (EAT - 26)
* Co-inhabiting with a study participant
* For former PORTIONS-3 study participants, when less than 3 months have passed since the last intervention visit (accepted if 3 or more months have elapsed).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy men and women living with overweight or obesity and willing to receive a 6-month intervention focused on changing their dietary habits
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2024-09-27 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in 24 h total dietary energy intake | Clinical investigation day 1 (week 0); Phone call (week 2, week 4, week 6, week 8, week 10); Clinical investigation day 2 (week 12); Phone call (week 14, week 16, week 18, week 20, week 22); Clinical investigation day 3 (week 24)
  24 h total dietary energy intake (in kcal) will be obtained from the 24 h dietary record
Change from baseline in 24 h total dietary volume intake | Clinical investigation day 1 (week 0); Phone call (week 2, week 4, week 6, week 8, week 10); Clinical investigation day 2 (week 12); Phone call (week 14, week 16, week 18, week 20, week 22); Clinical investigation day 3 (week 24)
  24 h total dietary volume intake (in g) will be obtained from the 24 h dietary record
Change from baseline in daily dietary energy density | Clinical investigation day 1 (week 0); Phone call (week 2, week 4, week 6, week 8, week 10); Clinical investigation day 2 (week 12); Phone call (week 14, week 16, week 18, week 20, week 22); Clinical investigation day 3 (week 24)
  24 h total dietary energy intake (kcal) and 24 h total dietary volumen intake (g) will be combined to report daily dietary energy density (in kcal/g). Daily dietary energy density is defined as the ratio of 24 h total dietary energy intake (in kcal) to the 24 h total dietary volume intake (in g)
Intervention adherence | Clinical investigation day 1 (week 0); Phone call (week 2, week 4, week 6, week 8, week 10); Clinical investigation day 2 (week 12); Phone call (week 14, week 16, week 18, week 20, week 22); Clinical investigation day 3 (week 24)
  Daily dietary energy density, meal nutrient composition and use of intervention components (spoon, oil dispenser, guide, app) will be combined to report intervention adherence (as a qualitative measure)

SECONDARY OUTCOMES:
Change from baseline in meal dietary energy density | Clinical investigation day 1 (week 0); Phone call (week 2, week 4, week 6, week 8, week 10); Clinical investigation day 2 (week 12); Phone call (week 14, week 16, week 18, week 20, week 22); Clinical investigation day 3 (week 24)
  Meal (breakfast, lunch and dinner) dietary energy density (kcal/g) will be calculated as the ratio of meal total dietary energy intake (in kcal) to the 24 h total dietary volume intake (in g), obtained from the 24 h dietary record
Change from baseline in meal nutrient composition: Grams | Clinical investigation day 1 (week 0); Phone call (week 2, week 4, week 6, week 8, week 10); Clinical investigation day 2 (week 12); Phone call (week 14, week 16, week 18, week 20, week 22); Clinical investigation day 3 (week 24)
  Meal (breakfast, lunch and dinner) nutrient content (in g) will be defined as the meal's content of carbohydrate (g), protein (g), vegetables (g), fibre (g), and sodium (mg) obtained from the 24 h dietary record
Change from baseline in meal nutrient composition: % energy | Clinical investigation day 1 (week 0); Phone call (week 2, week 4, week 6, week 8, week 10); Clinical investigation day 2 (week 12); Phone call (week 14, week 16, week 18, week 20, week 22); Clinical investigation day 3 (week 24)
  Percent of daily energy from meals will be defined as the % energy provided by carbohydrate, protein and vegetables at each meal (breakfast, lunch and dinner), obtained from the 24 h dietary record
Use of serving spoon (24 h frequency) | Phone call (week 2, week 4, week 6, week 8, week 10); Clinical investigation day 2 (week 12); Phone call (week 14, week 16, week 18, week 20, week 22); Clinical investigation day 3 (week 24)
  Number of times the intervention spoon has been used in a period of 24 h
Use of oil dispenser (24 h frequency) | Phone call (week 2, week 4, week 6, week 8, week 10); Clinical investigation day 2 (week 12); Phone call (week 14, week 16, week 18, week 20, week 22); Clinical investigation day 3 (week 24)
  Number of times the intervention oil dispenser has been used in a period of 24 h
Use of intervention guide (24 h frequency) | Phone call (week 2, week 4, week 6, week 8, week 10); Clinical investigation day 2 (week 12); Phone call (week 14, week 16, week 18, week 20, week 22); Clinical investigation day 3 (week 24)
  Number of times the intervention guide has been consulted in a period of 24 h
Use of intervention app (24 h frequency) | Phone call (week 14, week 16, week 18, week 20, week 22); Clinical investigation day 3 (week 24)
  Number of times the intervention app has been used in a period of 24 h
Use of serving spoon (15 day frequency) | Phone call (week 2, week 4, week 6, week 8, week 10); Clinical investigation day 2 (week 12); Phone call (week 14, week 16, week 18, week 20, week 22); Clinical investigation day 3 (week 24)
  Number of times the intervention spoon has been used in a period of 15 days
Use of oil dispenser (15 day frequency) | Phone call (week 2, week 4, week 6, week 8, week 10); Clinical investigation day 2 (week 12); Phone call (week 14, week 16, week 18, week 20, week 22); Clinical investigation day 3 (week 24)
  Number of times the intervention oil dispenser has been used in a period of 15 days
Use of intervention guide (15 day frequency) | Phone call (week 2, week 4, week 6, week 8, week 10); Clinical investigation day 2 (week 12); Phone call (week 14, week 16, week 18, week 20, week 22); Clinical investigation day 3 (week 24)
  Number of times the intervention guide has been consulted in a period of 15 days
Use of intervention app (15 day frequency) | Phone call (week 14, week 16, week 18, week 20, week 22); Clinical investigation day 3 (week 24)
  Number of times the intervention app has been used in a period of 15 days
Anthropometric profile: Change from baseline in Body Weight | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), clinical investigation day 3 (week 24)
  Weight will be measured in kg; Weight and height will be combined to report BMI in kg/m^2
Anthropometric profile: Body Height | Clinical investigation day 1 (week 0)
  Height will be measured in m using a stadiometer; Weight and height will be combined to report BMI in kg/m^2
Anthropometric profile: Change from baseline in Body Mass Index | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), clinical investigation day 3 (week 24)
  Weight and height will be combined to report BMI in kg/m^2
Anthropometric profile: Change from baseline in Waist circumference | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), clinical investigation day 3 (week 24)
  Waist circumference will be measured in cm using a measuring tape. Waist circumference and hip circumference will be combined to report Waist-to-hip ratio.
Anthropometric profile: Hip circumference | Clinical investigation day 1 (week 0)
  Hip circumference will be measured in cm using a measuring tape. Waist circumference and hip circumference will be combined to report Waist-to-hip ratio.
Anthropometric profile: Change from baseline in Waist-to-hip ratio | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), clinical investigation day 3 (week 24)
  Waist circumference and hip circumference will be combined to report Waist-to-hip ratio. Waist to hip ratio is defined as the ratio of the waist circumference (cm) to the hip circumference (cm)
Anthropometric profile: Change from baseline in body fat composition | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), clinical investigation day 3 (week 24)
  Body fat composition will be quantified as fat mass (in kg, %) from a body composition analyser
Biochemical profile: Change from baseline in fasting blood glucose | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), clinical investigation day 3 (week 24)
  Fasting blood glucose levels (mg/dL)
Biochemical profile: Change from baseline in fasting blood insulin | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), clinical investigation day 3 (week 24)
  Fasting blood insuliln levels (mIU/L)
Biochemical profile: Change from baseline in fasting blood triglycerides | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), clinical investigation day 3 (week 24)
  Fasting blood triglycerides levels (mg/dL)
Biochemical profile: Change from baseline in fasting blood cholesterol | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), clinical investigation day 3 (week 24)
  Fasting blood total cholesterol levels (mg/dL)
Biochemical profile: Change from baseline in fasting blood ghrelin | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), clinical investigation day 3 (week 24)
  Fasting blood total ghrelin levels (pg/mL)
Biochemical profile: Change from baseline in fasting blood leptin | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), clinical investigation day 3 (week 24)
  Fasting blood leptin levels (ng/mL)
Meal eating behaviour: Change from baseline in Eating rate | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), clinical investigation day 3 (week 24)
  Average amount of milkshake consumed per unit of time (g/min), based on validated methodology (Yeomans, 2000)
Meal eating behaviour: Change from baseline in bite size | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), clinical investigation day 3 (week 24)
  Average amount of milkshake consumed at each sip (g), based on validated methodology (Yeomans, 2000)
Meal eating behaviour: Change from baseline in meal duration | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), clinical investigation day 3 (week 24)
  Average time used to drink a milkshake (min), based on validated methodology (Yeomans, 2000)
Meal eating behaviour: Change from baseline in deceleration rate | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), clinical investigation day 3 (week 24)
  Average change in eating rate (g/sec-squared), based on validated methodology (Yeomans, 2000)
Inhibitory control pattern: Change from baseline in N200 wave latency | Clinical investigation day 1 (week 0), clinical investigation day 3 (week 24)
  N200 wave latency (milisec), based on the Go/No Go paradigm (Ochner et al., 2009)
Inhibitory control pattern: Change from baseline in N200 wave length | Clinical investigation day 1 (week 0), clinical investigation day 3 (week 24)
  N200 wave length (microV), based on the Go/No Go paradigm (Ochner et al., 2009)
Inhibitory control pattern: Change from baseline in P300 wave latency | Clinical investigation day 1 (week 0), clinical investigation day 3 (week 24)
  P300 wave latency (milisec), based on the Go/No Go paradigm (Ochner et al., 2009)
Inhibitory control pattern: Change from baseline in P300 wave length | Clinical investigation day 1 (week 0), clinical investigation day 3 (week 24)
  P300 wave length (microV), based on the Go/No Go paradigm (Ochner et al., 2009)
Learning task: Change from baseline in learned meal portion size | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), clinical investigation day 3 (week 24)
  % error in chosen portion sizes for starch, protein and vegetables of a virtual meal vs recommended portion sizes (based on Brunstrom & Rogers, 2009)
Learning task: Change from baseline in learned meal nutrient content | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), clinical investigation day 3 (week 24)
  % error in chosen nutrient content of a virtual meal vs recommended nutrient content (based on Brunstrom & Rogers, 2009)

OTHER OUTCOMES:
Socio-demographic and lifestyle data | Pre-screening
  Socio-demographic characteristics of the sample collected via self-reported questionnaire (age, sex, education, marital status, household composition, employment, physical activity level, smoking, alcohol intake)
Eating habits: Risk of eating disorders | Pre-screening
  Score in the Eating Attitudes Test-26, ranging from 0-78 points, validated by Garner et al., 1982. Scores above 20 suggest risk for presence of potential eating disorders.
Eating habits: Eating habits profile | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), clinical investigation day 3 (week 24)
  Profile defined by the combined Restraint (0-21 points), Disihnibition (0-16 points) and Susceptibilty to hunger (0-14 points) sub-scales scores of the Three Factor Eating Questionnaire (TFEQ), validated by Stunkard & Messick, 1985. Restraint values above 11, disinhibition values above 8 and susceptibility to hunger values above 4 are considered worse outcomes (i.e. risk for development of obesity and other eating disorders)
Eating habits: Portion control tool usage | Clinical investigation day 3 (week 24)
  Previous usage of portion control tools (end of study interview)
Eating habits: Frequency of home made meals | Pre-screening
  Frequency of consuming home made meals via self-reported questionnaire
Eating habits: Frequency of take away meals | Pre-screening
  Frequency of consuming take away meals via self-reported questionnaire
Eating habits: Meal prep and serving | Pre-screening
  Responsible person for cooking at home, via self-reported questionnaire
Eating habits: Liking for the intervention food (milkshake) | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), clinical investigation day 3 (week 24)
  Liking for the foods to be used in the intervention, via self-reported questionnaire (100 mm visual analogue scale)
Eating habits: Familiarity with the intervention food (milkshake) | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), clinical investigation day 3 (week 24)
  Familiarity with the foods to be used in the intervention, via self-reported questionnaire (100 mm visual analogue scale)
Eating habits: Appetite levels | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), clinical investigation day 3 (week 24)
  Scores for hunger, fullness, thirst, prospective intake, nausea measured on a 100 mm visual analogue scale before consumption of a milkshake (validated questionnaire based on Hill & Blundell, 1982)
Eating habits: Beverage consumption habits | Pre-screening (week 0), clinical investigation day 3 (week 24)
  Self-reported questionnaire assessing caloric beverage intake, awareness of beverage portion sizes and acceptance of portioning tools for liquids currently on the market (pre-piloted on-line BPS survey, Vargas-Alvarez et al., 2021)
Eating habits: Problem eating behaviour questionnaire (PEBQ) | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), clinical investigation day 3 (week 24)
  Validated questionnaire (Carter & Jansen, 2012) used to identify eating patterns associated with the risk for obesity. It consists of 25 items answered on a 5-Pt intensity scale. The information collected can be used qualitatively, to identify problematic behaviors, or quantitatively by adding the direct scores. Scores greater than 50 suggest a moderate to high frequency of behaviors associated with obesity.
Medical history | Pre-screening (week 0)
  Self-reported questionnaire based on previous studies (Almiron-Roig et al., 2023) asking about special dietary needs, pregnancy, lactation, menopause, history of eating disorders, history of mental illness, incompatible medical conditions (e.g. cancer, diabetes, memory loss), regular medication including nutritional and other supplements
Anthropometric profile: General body composition | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), clinical investigation day 3 (week 24)
  Fat mass distribution (trunk, arms, legs), fat-free mass (kg, %), fat-free mass distribution, basal metabolic rate (kcal/day)
Psychological profile: Personality | Pre-screening
  Score in the NEO-Five Factor Inventory (NEO-FFI) 60 item validated questionnaire (Costa & McCrae, 1989). The score for each central domain of normal personality defined by the Five-Factor Model of personality (neuroticism, extraversion, conscientiousness, agreeableness, and openness to experience) is calculated. A higher score on a scale assessing a certain personality domain indicates a stronger expression of traits associated with this particular domain
Psychological profile: Perceived stress | Pre-screening
  Score in the Perceived Stress Scale-14 (PSS-14) validated questionnaire (Cohen et al., 1983). Scores ranging from 0 to 13 suggest low stress, scores ranging from 14 to 24 suggest moderate stress, and scores above 27 suggest high perceived stress
Psychological profile: Emotional intelligence | Pre-screening
  Score in the Trait Meta-Mood Scale-24 (TMMS-24) validated questionnaire (Salovey et al., 1995). The score for three different dimensions of emotional intelligence are calculated. To obtain a score for each factor, items 1 to 8 are added for the emotional attention factor, items 9 to 16 for the emotional clarity factor, and items 17 to 24 for the emotional repair factor.
Psychological profile: Mood | Pre-screening
  Score in the Profile of Mood States (POMS) validated questionnaire (McNair et al., 1971). The score for six different dimensions of mood (tension, anger, fatigue, depression, confusion, and vigour) is calculated. A higher score on a scale assessing a certain mood dimension indicates a stronger expression of associated feelings. The resulting scores will range from -24 to 177, with lower scores indicative of people with more stable mood profiles
Attitude towards intervention: Intervention expectations | Clinical investigation day 1 (week 0)
  Self-constructed scale evaluated with the sum of scores (1-10) for 5 items (based on Nau & Borkovec, 1972). The 5 items include rating the intervention's logic, satisfaction, recommendability, expected usefulness, and the respondent's readiness to follow it. A higher score reflects a more positive expectation towards the upcoming intervention.
Attitude towards intervention: Intervention opinion | Clinical investigation day 2 (week 12), Clinical investigation day 3 (week 24)
  Self-constructed scale evaluated with the sum of scores (1-10) for 5 items (based on Nau & Borkovec, 1972). The 5 items include rating the intervention's logic, satisfaction, recommendability, usefulness, and the respondent's readiness/intention to continue with it. A higher score reflects a more positive opinion towards the experienced intervention.
Attitude towards intervention: Dietetic tool acceptance (serving spoon, oil dispenser) | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), Clinical investigation day 3 (week 24)
  Previously piloted questionnaire (Almiron-Roig et al., 2016) including 5-Pt Likert scores for portion tool attractiveness, fits within lifestyle, embarrassment, ease of use, perceived effectiveness and resistant to use. An average score of 1 or 2 indicates low acceptance, 3 neutral, and 4 or 5 high acceptance.
Attitude towards intervention: Intervention component acceptance (serving spoon, oil dispenser, intervention guide, intervention app) | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), Clinical investigation day 3 (week 24)
  Single scale instrument measuring the level of intention to use each component from 0-100 on a 100 mm visual analogue scale (previously piloted questionnaire, Almiron-Roig et al., 2016).
Attitude towards intervention: Perceived app usability | Clinical investigation day 2 (week 12), Clinical investigation day 3 (week 24)
  System Usability Scale (SUS) (based on Brooke, 1996). Includes ten 5-Pt Likert questions of which 5 items are scored positively (pleasant, easy to use, good functionality, quick to learn, safe), and 5 items are scored reversedly (complex, requires support, inconsistent, complicated to use, requires learning). A higher overall score indicates higher perceived usability.
Attitude towards intervention: Intervention guide assessment | Clinical investigation day 2 (week 12)
  Self-constructed questionnaire including 20 items answered with a 5-Pt Likert scale. The first 10 items assess content of the guide (credibility, coherence, usefulness, applicability) and the second 10 items assess format (organisation, word choice and communication style). A score <60 indicates poor assessment (the tool cannot be used in clinical practice as it stands); a score between 60-79 indicates the tool needs revision before implementation; a score of 80 or above indicates the tool is well rated by potential users and may be useful in clinical practice.
Intervention component usage: serving spoon | Phone call (week 2, week 4, week 6, week 8, week 10); Clinical investigation day 2 (week 12); Phone call (week 14, week 16, week 18, week 20, week 22); Clinical investigation day 3 (week 24)
  Types of meals in which the serving spoons were most frequently used
Intervention component usage: oil dispenser | Phone call (week 2, week 4, week 6, week 8, week 10); Clinical investigation day 2 (week 12); Phone call (week 14, week 16, week 18, week 20, week 22); Clinical investigation day 3 (week 24)
  Types of meals in which the oil dispenser was most frequently used
Intervention component usage: intervention guide | Phone call (week 2, week 4, week 6, week 8, week 10); Clinical investigation day 2 (week 12); Phone call (week 14, week 16, week 18, week 20, week 22); Clinical investigation day 3 (week 24)
  Guide sections most frequently checked
Intervention component usage: intervention app | Phone call (week 2, week 4, week 6, week 8, week 10); Clinical investigation day 2 (week 12); Phone call (week 14, week 16, week 18, week 20, week 22); Clinical investigation day 3 (week 24)
  App functions most frequently used
Protocol compliance on clinical investigation days | Clinical investigation day 1 (week 0), Clinical investigation day 2 (week 12), Clinical investigation day 3 (week 24)
  Self-constructed interview to verify participants' compliance with arrival time, physical activity and dietary requirements and any change in medication occurred prior to each clinical investigation day
End of study survey | Clinical investigation day 3 (week 24)
  Self-constructed interview to assess participant's overall experience with the intervention at study end (items include previous tools/methods employed, satisfaction with intervention, consistency of use, barriers experienced and intention to continue using the components)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Almiron-Roig, PhD, Principal Investigator — University of Navarra
Locations (1):
- University of Navarra, Dept. of Food Science and Physiology, Center for Nutrition Research, Pamplona, Navarre, Spain